CLINICAL TRIAL: NCT03758703
Title: Investigating Music Care Intervention On Palliative Care Patients
Brief Title: Music Intervention on Palliative Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Arbaaz Patel, Bachelor of Health Sciences Student at McMaster University, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5316
Record Dates: First submitted 2018-11-23; First posted 2018-11-29 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Palliative Care

STUDY DESIGN:
Intervention Model Description: This study will employ a pragmatic parallel randomized-control trial design as a mixed-methods study in which approximately half of the participants will be randomized into a control and the other remaining half in the experimental group.
Masking Description: Because of the nature of the intervention, it is not possible to perform blinding/masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-recorded music intervention group (Experimental): The experimental group will be receiving the pre-recorded music care intervention. The intervention is to be delivered once a day for 30 minutes, over one week, on a portable Bluetooth speaker system. Participants will select their own music from the list of pre-recorded songs playlist and are free to switch to another playlist within their treatment arm should they desire. This music was specifically designed for use in palliative care. Specifically, all songs are played at 60 beats per minute to mimic resting heart rate. Instrumentation was specifically chosen to be soothing and calming
  Interventions: Other: Pre-recorded music intervention group
- Pre-recorded soothing poetry group (Active Comparator): The control group will be provided pre-recorded soothing poetry which they will self-select. Participants are allowed to switch playlists within their treatment arm each day should they desire. This control group is designed to control time, attention, and placebo effect. Thus, the soothing poetry will be offered the identical time duration of listening to recorded soothing poetry readings and played at the same time the intervention group receives the pre-recorded music.
  Interventions: Other: Pre-recorded soothing poetry group

INTERVENTIONS:
Other: Pre-recorded music intervention group — Refer to the arm/group descriptions.
  Arms: Pre-recorded music intervention group
Other: Pre-recorded soothing poetry group — Refer to the arm/group descriptions.
  Arms: Pre-recorded soothing poetry group

SUMMARY:
Palliative/hospice care patients experience many negative symptoms during their time in such facilities. These symptoms include, but are usually not limited to, pain, anxiety, depression, and so on. This study is interested in exploring how a music intervention can be used to reduce these symptoms in order to improve the quality of life for these patients. Specifically, because music interventions can be costly (e.g., employing music therapists and the likes of) and there is a lack of knowledge about how to properly implement music interventions, we believe that it would be most cost-effective as well as effective in reducing the described symptoms by introducing pre-recorded music as an intervention. Patients will be given pre-recorded music which requires less training and less money but may be just as effective as music interventions that do not use pre-recorded music. Patients will be evaluated by administering surveys at predetermined times to measure their symptoms, and interview-like questions will be administered at the end of the study to collect information that will be used to inform a larger study in the future. This study will, therefore, be collecting data on both how effective the intervention is and how feasible it is to use the same methods for a similar larger study in the future.

DETAILED DESCRIPTION:
This study will employ a pragmatic randomized control trial design as a mixed-methods study in which approximately half of the participants will be randomized into a control and the other remaining half in the experimental group. Randomization sequences will be generated externally and allocation concealment will be employed. Group allocation will be revealed to subjects following informed consent, which is characterized by participants understanding the full details of this study and any risks that may present themselves. Because of the nature of the intervention, it is not possible to perform blinding and further stratification is restricted due to the small sample size. Confounding variables, like those of age, gender, education, and cancer-type, will be collected and controlled for during the statistical analyses. In addition, palliative performance status (PPS) at baseline, and daily pain medication usage during the intervention will be recorded to control for potential confounders. PPS is regularly measured by hospital staff. The research team will not access the resident's health records. Instead, the in-house care staff will perform this screening and refer eligible participants to the research team. Participants randomized into the experimental group will receive and self-select a pre-recorded music care playlist, whereas those randomized into the control group will receive and self-select a pre-recorded soothing poetry playlist, daily, over the course of seven days, but are free to select different playlists within their intervention arm each day. The music and poetry will be delivered using the same system with the same sound quality through a portable Bluetooth speaker system. The speaker system will allow others to listen with the participant. Pre-recorded poetry was chosen as a control intervention because it stimulates the same biological auditory system as music. This is an appropriate comparison for the pre-recorded music intervention because although it is delivered through the same fundamental biological pathway, poetry sound waves are interpreted as non-patterned and non-musical. In contrast, music sound waves are interpreted as patterned and organized. It is important to recognize that, especially in the context of hospice care, it would be unethical to prevent participants from using music outside of the study. This is controlled for by performing pre- and post-evaluations exclusively for the session. In other words, this data will be collected concurrently rather than longitudinally. Further, an additional daily involvement questionnaire will be used to determine whether music has been used outside of the context of this study. This will allow the research team to later control for this (e.g., when it is used as a distraction technique outside of this study). At the end of each intervention, which will last for 30-minutes, three validated questionnaires (hospice quality of life index-revised (HQLIR), stait-trait anxiety inventory scale (STAIS), and edmonton symptom assessment scale (ESAS)) will be administered in order to evaluate the effectiveness of the intervention. However, one of these questionnaires will only be administered on day one, three, and seven. Finally, an additional "daily involvement" questionnaire will be used as a means to ensure that the music intervention took place. This questionnaire will be completed on each of the seven days for each participant and will record their daily involvement. The individual administering the above-mentioned questionnaires will remain with the resident for the duration of the intervention and listen to the intervention together with the resident; this holds true for both the control and experimental group. At the end of the study, acceptability data measuring trial feasibility as a function of recruitment process; participation/refusal rate; study measurements completion rate; and protocol adherence including intervention delivery and data collection, will be collected via audio-recorded semi-structured interviews with residents, families, and healthcare providers/volunteers for which consent will first be collected. Resident's families will be invited by the participant for involvement in processes such as listening to the intervention with the resident or being present during the questionnaire process, and will be given the opportunity to consent prior to engaging in the semi-structured interview. All above-mentioned questionnaires will be administered by either community volunteers, study investigators, and/or hospice staff. Note that all questionnaires will be de-identified. In order to correctly code questionnaires based on each participant's unique study identifier, first and last names will be recorded for each participant upon enrolment in the study. First and last names will be recorded on the hard-copy study code sheet which will be kept in the PI's locked filing cabinet. The code sheet will be used to prepare the de-identified questionnaires which will be used to collect data in the community hospices. Upon completion of the study, the hard copy code sheet will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking;
* A score of 3 or higher on ESAS scale for pain and anxiety
* Cognitively alert and competent to provide informed consent
* A Palliative Performance Scale of at least 40/100.

Exclusion Criteria:

* Participants with a prognosis of fewer than 2 weeks or an expectation of leaving the inpatient setting within a 2 week period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Assessing changes in quality of life in palliative care patients | 3 days (days 1,3 and 7 of data collection)
  Self-report Hospice Quality of Life Index-Revised (HQLI-R) questionnaire with 29 items; each question ranges from 0 to 10 (0 indicating the lowest quality and 10 indicating the highest quality). This yields a total score between 0 and 290.
Assessing changes in symptom severity in palliative care patients | 7 days (days 1 through 7 of data collection)
  Self-report Edmonton Symptom Assessment Scale-revised (ESAS-R) questionnaire with 10 items; each item ranges from 0 to 10 (0 indicating low to no severity in symptoms or that the symptom is absent, and 10 indicating the highest symptom severity). This yields a total score between 0 and 100.
Assessing changes in trait and state anxiety in palliative care patients | 7 days (days 1 through 7 of data collection)
  Self-report State-Trait Anxiety Inventory Scale (STAI-S) questionnaire with 20 items; each item ranges from 1 to 4 (1 indicating low to no anxiety and 4 indicating the highest anxiety). This yields a total score between 0 and 80.

SECONDARY OUTCOMES:
Assessing trial feasibility for a larger future RCT | 1 day (day 7 of data collection)
  Trial feasibility will be collected in the form of audio-recorded semi-structured interviews to ascertain the feasibility of the method and logistics of the intervention. This knowledge will be applied to a future RCT in order to deliver the intervention more effectively and improve the data collection process.

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Mackinnon, MA, MMIE, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Emmanuel House Good Shepherd Residential Hospice, Hamilton, Ontario
  - Dr Bob Kemp Hospice, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
Only anonymized grouped data will be shared for publication once data analysis is complete.

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Care at the End of Life; Field MJ, Cassel CK, editors. Approaching Death: Improving Care at the End of Life. Washington (DC): National Academies Press (US); 1997. Available from http://www.ncbi.nlm.nih.gov/books/NBK233605/ PMID 25121204
- [Background] Morrison RS, Meier DE. Clinical practice. Palliative care. N Engl J Med. 2004 Jun 17;350(25):2582-90. doi: 10.1056/NEJMcp035232. No abstract available. PMID 15201415
- [Background] O'Callaghan CC. Pain, music creativity and music therapy in palliative care. Am J Hosp Palliat Care. 1996 Mar-Apr;13(2):43-9. doi: 10.1177/104990919601300211. PMID 8716327
- [Background] Archie P, Bruera E, Cohen L. Music-based interventions in palliative cancer care: a review of quantitative studies and neurobiological literature. Support Care Cancer. 2013 Sep;21(9):2609-24. doi: 10.1007/s00520-013-1841-4. Epub 2013 May 30. PMID 23715815
- [Background] Clements-Cortes A. The use of music in facilitating emotional expression in the terminally ill. Am J Hosp Palliat Care. 2004 Jul-Aug;21(4):255-60. doi: 10.1177/104990910402100406. PMID 15315187
- [Background] Olofsson A, Fossum B. Perspectives on music therapy in adult cancer care: a hermeneutic study. Oncol Nurs Forum. 2009 Jul;36(4):E223-31. doi: 10.1188/09.ONF.E223-E231. PMID 19581226
- [Background] Bradt J, Dileo C, Magill L, Teague A. Music interventions for improving psychological and physical outcomes in cancer patients. Cochrane Database Syst Rev. 2016 Aug 15;(8):CD006911. doi: 10.1002/14651858.CD006911.pub3. PMID 27524661
- [Background] McMillan SC, Weitzner M. Quality of life in cancer patients: use of a revised Hospice Index. Cancer Pract. 1998 Sep-Oct;6(5):282-8. doi: 10.1046/j.1523-5394.1998.00023.x. PMID 9767348
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Background] Spielberger CD, Gorsuch RL, Lushene R, Vagg PR, Jacobs GA. Manual for the state-trait anxiety inventory (Palo Alto, CA, Consulting Psychologists Press). Inc. 1983.
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Abbott JH. The distinction between randomized clinical trials (RCTs) and preliminary feasibility and pilot studies: what they are and are not. J Orthop Sports Phys Ther. 2014 Aug;44(8):555-8. doi: 10.2519/jospt.2014.0110. No abstract available. PMID 25082389
- See also: The State of Seniors Health Care in Canada — https://www.cma.ca/sites/default/files/2018-11/the-state-of-seniors-health-care-in-canada-september-2016.pdf
- See also: What Canadians Say: The Way Forward Survey Report — http://www.hpcintegration.ca/media/51032/The%20Way%20Forward%20-%20What%20Canadians%20Say%20-%20Survey%20Report%20Final%20Dec%202013.pdf
- See also: Episodes of Relationship Completion Through Song in Palliative Care — https://tspace.library.utoronto.ca/handle/1807/17744